CLINICAL TRIAL: NCT01493349
Title: The Role of Intestinal Microbiota Composition and Intestinal Permeability in the Development of (Complicated) Diverticular Disease.
Brief Title: Pathophysiology of Diverticular Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-2-058
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Colonic Diverticula; Diverticulitis
Keywords: Colonic diverticula; Diverticulitis
MeSH Terms: conditions — Diverticulum, Colon; Diverticulitis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — * 1 bloodsample (14.5mL)
  * 9 Colonic mucosal biopsies
  * 1 Intestinal washing sample (at least 15mL)
  * 1 Fecal sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Controls: No diverticular disease or other gastrointestinal and liver diseases
- Uncomplicated diverticular disease
- History of complicated diverticular disease
- Current complicated diverticular disease

SUMMARY:
Colonic diverticular disease is a highly prevalent condition in Western populations. The prevalence increases age-dependently from 5% at 40 years to 65% by the age of 85 years (1-3). The majority remain asymptomatic. However, a significant proportion of the patient population develops complications, such as diverticulitis with or without symptoms (10-20%) (1, 4-10). Perforated diverticulitis is rare with an estimated incidence of 4 per 100.000 per year, but the associated mortality rate is 22% to 39% (9, 11, 12). In the United States, the complications related to diverticular disease account for 130.000 hospitalizations each year, resulting in substantial health care costs (13). In Europe, it is estimated that approximately 23.600 deaths per year can be attributed to complicated diverticular disease, and the mortality will probably increase in the future due to the aging population (15-17). Several case studies report an overall increase in the incidence of diverticulitis, based on the increase in hospitalizations (18). Kang et al, reported a 16% increased male admission rate and 12% female admission rate for diverticulitis, between 1989/1990 and 1999/2000 (19). Aging and the Western diet, low in fiber and high in fat, in combination with increased intraluminal pressure and alterations in colonic motility are considered important etiological factors. A disturbance in large bowel motility is suggested to be a common pathophysiological feature in IBS and diverticular disease (20, 21). Based on observations that IBD, subgroups of IBS and (symptomatic) diverticular disease share clinical symptoms, the hypothesis is derived that they might also share pathophysiological factors like low grade inflammation, changed microbiota composition and activity, and increased intestinal permeability. The identification of clinical and pathophysiological factors associated with an increased risk for complicated diverticular disease may help to identify patients with diverticular disease, prevent complications, develop strategies to improve quality of life and reduce the related health care costs. Therefore we aim to investigate the composition of luminal and mucosal intestinal microbiota and the intestinal permeability in the development of diverticular disease and complicated diverticular disease. We hypothesize that both the intestinal microbiota and intestinal permeability are altered in patients with (current- or previous history of complicated) diverticular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years and ≤ 75 years
* Scheduled for colonoscopy
* Written informed consent
* Patient group: The presence of diverticulosis, diagnosed during the scheduled colonoscopy
* Control group: During the scheduled colonoscopy, diverticulosis or other
* gastrointestinal and liver diseases are absent. In other words, the
* colonoscopy is qualified as a 'normal' colonoscopy.

Exclusion Criteria:

* Age < 18 years
* Presence of gastrointestinal and liver diseases, such as inflammatory bowel disease.
* Use of NSAID's and proton pump inhibitors, during the 5-day time period prior to endoscopy.
* Alcohol intake above 14 consumptions per week for males and 7 consumption per week for females
* (Sub)total colectomy or hemicolectomy.
* Refusal to participate in this study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the hospital by their general practitioner
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
intestinal (luminal and mucosal) microbiota composition | up to 2 years

SECONDARY OUTCOMES:
Expression of tight junction proteins | up to 2 years
Intestinal permeability | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: A. M. Masclee, MD, PhD, Principal Investigator — Maastricht University Medical Center; D. Jonkers, PhD, Study Chair — Maastricht University Medical Center; R. C. Deutz, MD, Study Chair — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands